CLINICAL TRIAL: NCT01889264
Title: Methionine Metabolism in Enterally Fed Critically Ill Children
Brief Title: Methionine Metabolism in Enterally Fed Pediatric Sepsis
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Leticia Castillo, Department Chair Peds Critical Care, The Cleveland Clinic
Other Study IDs: STU-042011-088
Record Dates: First submitted 2013-05-24; First posted 2013-06-28 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Sepsis; Critical Illness
Keywords: Methionine Metabolism; Enteral Nutrition; Pediatric; Pediatrics; Sepsis; Observational Study
MeSH Terms: conditions — Sepsis; Critical Illness | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critically Ill Pediatric Patients: Critically ill septic pediatric patients, Age 1 month-3 years, Age 4-12 years and Age 13-19 years, males and females
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational, Translational non-treatment study

SUMMARY:
Critically ill children have abnormal utilization of nutrients such as glucose, lipids and protein. Protein synthesis is increased mainly in the form of immune and signaling proteins, while muscle and structural protein synthesis is decreased. The metabolism of sulfur amino acids through the splanchnic area and specifically methionine and cysteine have not been investigated in critically ill septic children, despite that sulfur amino acids have important roles in thiol, antioxidant and epigenetic reactions. Methionine metabolism in sick children will be influenced by its rate of utilization through different pathways. Our study aims to investigate the metabolism of methionine and cysteine when both amino acids are given by the enteral route in critically ill septic children. The investigators are focused on the rates of transmethylation, remethylation and transsulfuration in critically ill septic children, and if the current standard nutrition maintains methionine nutritional balance and functional requirements in critically ill children fed by the enteral route.

DETAILED DESCRIPTION:
This is a prospective, translational study on the splanchnic metabolism of methionine to determine the rates of the different pathways and synthesis rates of glutathione when critically ill children are fed by the enteral route, and the difference among various age groups. The study size will include 45 critically ill septic, pediatric patients (15 infants at 1 month-3 years of age, 15 children at 4-12 years of age and 15 adolescent at 13-19 years of age), males and females admitted to the pediatric intensive care unit (PICU) at Children's Medical Center, Dallas. The minimal subject's weight will be 4 kg. The number of subjects includes an expected drop out rate of about 20%, in order to obtain 15 patients with complete data in each group. Patients will receive nutritional support as per standard care. This study will yield important knowledge and may lead in the future to changes in the current practice on the management of critically ill pediatric patients in the PICU.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 1 month-19 years
2. Diagnosis of severe sepsis diagnosed as clinical sepsis syndrome (requires two of the following criteria):

   * Source of infection
   * Fever or Hypothermia
   * Leukocytosis or Leucopenia
   * Poor organ perfusion (such as delayed capillary refill or decreased urine output or hypotension)
   * Bacteremic sepsis demonstrated by positive blood culture
3. Weight greater or equal to 4.0 kg
4. Need for enteral nutrition by a nasogastric/nasoduodenal tube
5. Presence of central and/or arterial venous access as per clinical indication

Exclusion Criteria:

1. Patients with metabolic diseases (i.e. Insulin dependent diabetes mellitus, urea cycle disorders, cystinuria, etc.)
2. Pregnancy
3. Primary liver failure
4. Primary renal failure
5. Patients unable to tolerate enteral feedings
6. Weight less than 4.0 kg

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Septic pediatric patients: A total of 45 critically ill children age 1 month-19 years with diagnosis of sepsis, as defined by the International Sepsis Consensus Conference.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Methionine Metabolism | Clinical Signs, AEs, SAEs, CO2, Tracer Infusion, Blood: (Baseline - 8 hours)
  Rates of transmethylation, remethylation and transsulfuration and erythrocyte GSH synthesis when nutrients are given by the enteral route in pediatric critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Castillo, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States